CLINICAL TRIAL: NCT03060980
Title: A Phase 3b, Randomized, Active Comparator, Open-label, Multicenter Study to Compare the Efficacy, Safety, and Tolerability of ITCA 650 to Empagliflozin and to Glimepiride as Add-on Therapy to Metformin in Patients With Type 2 Diabetes
Brief Title: Comparison of Efficacy, Safety, and Tolerability of ITCA 650 to Empagliflozin and Glimepiride as add-on Metformin
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Decision by Sponsor
Sponsor: Intarcia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITCA 650-CLP-203
Record Dates: First submitted 2017-02-09; First posted 2017-02-23 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide; empagliflozin; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Experimental: Group 1 (Experimental): ITCA 650 20/60 mcg/day
  Interventions: Drug: ITCA 650 20/60 mcg/day
- Experimental: Group 2 (Experimental): Empagliflozin 10 mg/day and 25 mg/day
  Interventions: Drug: Empagliflozin (oral)
- Experimental: Group 3 (Experimental): Glimepiride 1-6 mg/day
  Interventions: Drug: Glimepiride (oral)

INTERVENTIONS:
Drug: ITCA 650 20/60 mcg/day — ITCA 650 osmotic mini-pump delivering exenatide 20/60 mcg/day
  Arms: Experimental: Group 1
Drug: Empagliflozin (oral) — 10 mg/day and 25 mg/day
  Arms: Experimental: Group 2
Drug: Glimepiride (oral) — 1-6 mg/day
  Arms: Experimental: Group 3

SUMMARY:
A Phase 3b, open-label, randomized, multicenter, efficacy, safety, and tolerability study of ITCA 650 compared to Empagliflozin and to Glimepiride, as add-on therapy to Metformin in patients with Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2D 3 months prior to the Screening Visit.
* Body mass index (BMI) between ≥25 to ≤45 kg/m2 at the Screening Visit.
* Glycosylated hemoglobin A1c (HbA1c) ≥7.5 and ≤10.5%. 5. 6. On a stable (3 months prior to the Screening Visit) treatment regimen of metformin monotherapy of ≥1500 mg/day).

Exclusion Criteria:

* History of type 1 diabetes.
* Prior participation in a clinical study involving ITCA 650.
* Treatment with any GLP-1 receptor agonist (eg, liraglutide, exenatide) within 6 months prior to Screening.
* History or evidence, within the last 6 months prior to the Screening Visit, of myocardial infarction, coronary revascularization (coronary artery bypass grafting or percutaneous coronary intervention), unstable angina, or cerebrovascular accident or stroke.
* History or evidence of acute or chronic pancreatitis.
* History of medullary thyroid cancer or a family or personal history of multiple endocrine neoplasia type 2.
* Treatment of medications that affect GI motility.
* History of hypersensitivity to exenatide, empagliflozin, or glimepiride or to one of its excipients.
* Women that are pregnant, lactating, or planning to become pregnant.
* Chronic (>10 consecutive days) treatment with systemic corticosteroids within 8 weeks prior to screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2018-01-26 (Actual)

PRIMARY OUTCOMES:
Reduction in glycosylated hemoglobin A1c | Randomization to 69 weeks
  To determine whether ITCA 650 is non-inferior either to empagliflozin or to glimepiride in reducing glycosylated hemoglobin A1c (HbA1c) in patients with T2D following 65 weeks of treatment and 4 weeks of post treatment follow up.
Reduction in weight | Randomization to 69 weeks
  To determine whether ITCA 650 is non-inferior either to empagliflozin or to glimepiride in reducing weight in patients with T2D following 65 weeks of treatment and 4 weeks of post treatment follow up.

CONTACTS AND LOCATIONS:
Locations (100):
- United States (95):
  - Fountain Hills Family Practice, P.C., Fountain Hills, Arizona
  - Thomas C. Lenzmeier, M.D., P.C., Glendale, Arizona
  - Family Practice Specialists, Phoenix, Arizona
  - Central Phoenix Medical Center, Phoenix, Arizona
  - Fiel Family and Sports Medicine, Tempe, Arizona
  - Arizona Community Physicians, Tucson, Arizona
  - Orange Grove Family Practice, Tucson, Arizona
  - Anaheim Clinical Trials, Anaheim, California
  - Radiant Research, Carlsbad, California
  - Research Center of Fresno, Inc., Fresno, California
  - Marin Endocrine Care and Research, Inc., Greenbrae, California
  - National Research Institute, Huntington Park, California
  - National Research Institute, Los Angeles, California
  - Catalina Research Institute, Montclair, California
  - Providence Clinical Research, North Hollywood, California
  - Center for Clinical Trials of Sacramento, Inc., Sacramento, California
  - Denver VA Medical Center, Aurora, Colorado
  - Radiant Research, Centennial, Colorado
  - Colorado Springs Health Partners - East, Colorado Springs, Colorado
  - Columbine Family Practice, Littleton, Colorado
  - Nature Coast Clinical Reseaerch - Crystal River, Crystal River, Florida
  - Indago Research and Health Center, Inc., Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Research Institure of South Florida, Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Palm Harbor Medical Associates, Palm Harbor, Florida
  - Andres Patron, D.O., P.A, Pembroke Pines, Florida
  - South Broward Research, Pembroke Pines, Florida
  - Primary Care Research Group, Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Solaris Clinical Research, Meridian, Idaho
  - Michigan Avenue Internists, Chicago, Illinois
  - Medical and Procedural Specialists, Skokie, Illinois
  - HSHS Medical Group DIabetes Research, Springfield, Illinois
  - Community Hospital of Anderson and Madison County, Inc., Anderson, Indiana
  - Clinical Research Advantage, Evansville, Indiana
  - American Health Network of Indiana, LLC, Franklin, Indiana
  - American Health Network of Indiana, LLC, New Albany, Indiana
  - Heartland Research Associates, LLC, Augusta, Kansas
  - Overland Park Surgical Specialists, LLL dba College Park Family Care Center, Overland Park, Kansas
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Maine Research Associates, Auburn, Maine
  - Joslin Diabetes Center, Boston, Massachusetts
  - Radiant Research, Inc., Edina, Minnesota
  - Ehrhardt Clinical Research, LLC, Belton, Missouri
  - HealthCare Research Network, Hazelwood, Missouri
  - Mercury Street Medical Group, Butte, Montana
  - Skyline Medical Center, Elkhorn, Nebraska
  - Nevada Family Care, Henderson, Nevada
  - Palm Research Center, Inc., Las Vegas, Nevada
  - Albany Medical College, Albany, New York
  - Scott Research Center, Laurelton, New York
  - American Health Research, Charlotte, North Carolina
  - Medication Management, LLC, Greensboro, North Carolina
  - Down East Medical Associates, PA, Morehead City, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Radiant Research, Akron, Ohio
  - Sentral Clinical Research Services, LLC, Cincinnati, Ohio
  - Canyon Medical Center, LLC, Columbus, Ohio
  - Aventiv Research, Columbus, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Wells Institute for Health Awareness, Kettering, Ohio
  - University of Toledo, Toledo, Ohio
  - Oklahoma City Clinic - Midwest City, Midwest City, Oklahoma
  - Intend Research, Norman, Oklahoma
  - Oklahoma City Clinic - Central, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Harleysville Medical Associates, Harleysville, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Preferred Primary Care Phys Inc, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Holston Medical Group, P.C., Kingsport, Tennessee
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - DCT-AACT, LLC dba Discovery Clinical Trials, Austin, Texas
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - Research Institute of Dallas, Dallas, Texas
  - Global Medical Research, DeSoto, Texas
  - Juno Research, Houston, Texas
  - PCP for Life - -Tidwell, Houston, Texas
  - Sante Clinical Research, Kerrville, Texas
  - Health Texas Research Institute, San Angelo, Texas
  - Panacea Clinical Research, San Antonio, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Victorium Clinical Research Ltd., San Antonio, Texas
  - MacGregor Medical Center, San Antonio, Texas
  - Crossroads Clinical Research, LLC, Victoria, Texas
  - Ericksen Research and Development, LLC, Clinton, Utah
  - Radiant Research, Murray, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - Sound Healthcare, Port Orchard, Washington
- Canada (5):
  - Bailey Clinic, Red Deer, Alberta
  - CookMed Research, Victoria, British Columbia
  - Milestone Research, London, Ontario
  - Bluewater Clinical Research Group, Sarnia, Ontario
  - Dr. Anil K. Gupta Medicine Professional Corporation, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No